CLINICAL TRIAL: NCT03036085
Title: Liposomal Bupivacaine Versus Bupivacaine for Postoperative Analgesia Following Video-assisted Thoracoscopic Surgery.
Brief Title: Liposomal Bupivacaine for Pain Control Following Thoracic Surgery.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Harald Ott, Associate Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016P002754
Record Dates: First submitted 2016-12-09; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Pain, Postoperative; Thoracic Diseases; Local Anesthetics Causing Adverse Effects in Therapeutic Use; Opioid Dependence
Keywords: postoperative pain; video-assisted thoracoscopic surgery (VATS); opioids; bupivacaine; liposomal bupivacaine; analgesia; local anesthetics
MeSH Terms: conditions — Pain, Postoperative; Thoracic Diseases; Opioid-Related Disorders; Agnosia | interventions — Bupivacaine; Epinephrine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine (Active Comparator): Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with 0.5% bupivacaine with 1% epinephrine. In the bupivacaine group 20 ml of 0.5% bupivacaine with 1% epinephrine will be diluted to a total volume of 40 ml using 20 ml normal saline. From those 40 ml, 30 ml will be used for the posterior intercostal nerve block and 10 ml will be injected locally into the surgical wounds.
  Interventions: Drug: Bupivacaine; Drug: Epinephrine; Drug: Normal saline
- Liposomal bupivacaine (Experimental): Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with liposomal bupivacaine (13.3 mg/ml). In the liposomal bupivacaine group, a total dose of 266 mg of liposomal bupivacaine (one 20 ml vial of 13.3 mg/ml) per patient will be diluted to a total volume of 40 ml using 20 ml normal saline.
  Interventions: Drug: Liposomal bupivacaine; Drug: Normal saline

INTERVENTIONS:
Drug: Liposomal bupivacaine — In the operating room after induction of general anesthesia patients will be positioned in a lateral decubitus position, prepared and draped in a sterile fashion. Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with liposomal bupivacaine plus normal saline.
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: Bupivacaine — In the operating room after induction of general anesthesia patients will be positioned in a lateral decubitus position, prepared and draped in a sterile fashion. Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with bupivacaine plus epinephrine plus normal saline.
  Other Names: Marcaine; Marcain; Sensorcaine; Vivacaine
  Arms: Bupivacaine
Drug: Epinephrine — In the operating room after induction of general anesthesia patients will be positioned in a lateral decubitus position, prepared and draped in a sterile fashion. Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with bupivacaine plus epinephrine plus normal saline.
  Other Names: Adrenaline; Adrenalin
  Arms: Bupivacaine
Drug: Normal saline — In the operating room after induction of general anesthesia patients will be positioned in a lateral decubitus position, prepared and draped in a sterile fashion. Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with liposomal bupivacaine plus normal saline or with bupivacaine plus epinephrine plus normal saline.

SUMMARY:
The aims of the study are to compare the effectiveness and postoperative outcomes of liposomal bupivacaine vs plain bupivacaine following video-assisted thoracoscopic surgery. The investigators' hypothesis is that liposomal bupivacaine will decrease the postoperative pain and will be associated with more favorable postoperative outcomes when compared to plain bupivacaine following video-assisted thoracoscopic surgery.

DETAILED DESCRIPTION:
Pain management remains a primary concern for many patients following thoracic surgery. Suboptimal analgesia leads to numerous postoperative complications like reduced cardiac, respiratory and gastrointestinal functions, more septic and thromboembolic complications, increased incidence of developing chronic pain states, increased mortality in high-risk patients with multiple comorbidities, and many others.

Opioids have a distinct role in the postoperative analgesia. Although opioids have positively affected surgery for decades, they are associated with a number of potentially severe side effects including prolonged ileus, nausea, vomiting, central nervous system and respiratory depression, development of hyperalgesia, and the risk of dependency and abuse. These adverse effects increase the overall cost of treatment for these patients and can potentially result in longer hospital stays.

Local infiltration and regional blocks of local anesthetics are increasingly utilized during thoracic surgery procedures as an alternative to epidural analgesia. Bupivacaine is widely used for intercostal nerve blocks but its utility is limited by its short duration of action (<6 hours). Perineural catheters for continuous infusion of bupivacaine have been used to overcome this limitation but the need of expensive pumps and the risk of significant complications associated with the use of catheters (i.e. infection, septicemia, intravascular migration etc) has limited its use.

Encapsulation of local anesthetics into liposomes is a novel method which extends drug delivery. The use of multivesicular liposomes has been shown to provide a slow and steady release of local anesthetics for several days after nonvascular administration. Liposomal bupivacaine is a novel formulary of bupivacaine, is designed for a single-dose local infiltration into the surgical site and produces postsurgical analgesia for up to 72-96 hours.

Liposomal bupivacaine is not currently licensed by the U.S. Food and Drug Administration for peripheral nerve block but has been approved for single-dose infiltration into the surgical site. However, it has been shown in two retrospective studies of patients with open thoracotomies for lung, pleural or mediastinal pathologies that liposomal bupivacaine intercostal nerve blockade is associated with increased pain control and decreased length of hospital stay compared to thoracic epidural analgesia.

This is a single-blind randomized prospective research study comparing pain control and postoperative outcomes following intercostal neural blockade with liposomal bupivacaine versus plain bupivacaine plus epinephrine during video-assisted thoracoscopic surgical procedures. Eligible patients would be all patients aged older than 18 years who undergo a video-assisted thoracoscopic lung resection at Massachusetts General Hospital. Pregnant women, prisoners, emergent cases, patients under 18 years, and patients with chronic pain, documented alcohol or drug abuse and allergies to bupivacaine will be excluded from this study.

Primary end point will be self-reported pain score on a visual analog scale from 0 to 10 at postoperative day #1. By utilizing a mean difference in self-reported pain scores of 1 point with a standard deviation of 2.5 points, a sample size of 100 patients per group would be needed for a power (beta) of 0.8 and probability level (alpha) of 0.05. All patients would be enrolled at Massachusetts General Hospital.

The video-assisted thoracoscopic surgeries and intercostal nerve blockade with plain bupivacaine plus epinephrine or liposomal bupivacaine will be performed by all thoracic surgeons at Massachusetts General Hospital. In the operating room after induction of general anesthesia patients will be positioned in a lateral decubitus position, prepared and draped in a sterile fashion. Under thoracoscopic guidance, a posterior intercostal nerve block will be performed with liposomal bupivacaine (13.3 mg/ml) or 0.5% bupivacaine with 1% epinephrine. In the liposomal bupivacaine group, a total dose of 266 mg of liposomal bupivacaine (one 20 ml vial of 13.3 mg/ml) per patient will be diluted to a total volume of 40 ml using 20 ml normal saline. In the bupivacaine group 20 ml of 0.5% bupivacaine with 1% epinephrine will be diluted to a total volume of 40 ml using 20 ml normal saline. From those 40 ml, 30 ml will be used for the posterior intercostal nerve block and 10 ml will be injected locally into the surgical wounds.

If immediate postoperative pain scores were rated 4/10 or greater, an intravenous patient controlled analgesia device will be provided with hydromorphone 0.2 mg every 10 minutes or nonopioid analgesics as needed. No narcotics will be given in the spinal space. Oral metoclopramide or ondansetron will be given as needed to combat the side effects of the narcotics.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients would be all patients aged older than 18 years who undergo a video-assisted thoracoscopic lung resection at Massachusetts General Hospital.

Exclusion Criteria:

* Pregnant women, prisoners, emergent cases, patients under 18 years, and patients with chronic pain, documented alcohol or drug abuse and allergies to bupivacaine will be excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patient self-reported pain visual analog scale score - Day 1 | Postoperative Day #1

SECONDARY OUTCOMES:
Patient self-reported pain visual analog scale score - Day 3 | Postoperative Day #3
Patient self-reported pain visual analog scale score - Discharge | At the day of discharge from the hospital. Discharge day could be on average postoperative day #4 or #5.
Time until first opioid usage | After the surgery and until the participant receives the first opioid medication, assessed up to 10 days after surgery.
Total opioid usage (in morphine equivalents) | After the surgery and until the participant is discharged from the hospital. Discharge day could be on average postoperative day #4 or #5.
Anti-emetic usage | After the surgery and until the participant is discharged from the hospital. Discharge day could be on average postoperative day #4 or #5.
Naloxone usage | After the surgery and until the participant is discharged from the hospital. Discharge day could be on average postoperative day #4 or #5.
Length of hospital stay | After the surgery and until the participant is discharged from the hospital. Discharge day could be on average postoperative day #4 or #5.
Postoperative complications (e.g. pneumonia, pulmonary complications, wound infections etc) | The first 30 days after surgery
Time to ambulation | After the surgery and until the participant starts ambulating during hospitalization, assessed up to 10 days after surgery.
Time to first bowel movement | After the surgery and until the participant has the first bowel movement during hospitalization, assessed up to 10 days after surgery.
Time to chest tube removal | After the surgery and until the participant has his/her chest tube removed during hospitalization, assessed up to 10 days after surgery.
Peak expiratory flow measurements | Measured twice daily following surgery until the participant is discharged from the hospital. Discharge day could be on average postoperative day #4 or #5.
  Measures air flowing in and out of the lungs.
Peak expiratory flow measurements | Measured twice daily the day at the first postoperative visit (usually within 10-30 days postoperatively)
  Measures air flowing in and out of the lungs.

CONTACTS AND LOCATIONS:
Overall Officials: Harald Ott, MD, Principal Investigator — Division of Thoracic Surgery, Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen AH. Toxicity and allergy to local anesthesia. J Calif Dent Assoc. 1998 Sep;26(9):683-92. PMID 9879238
- [Result] Apfelbaum JL, Chen C, Mehta SS, Gan TJ. Postoperative pain experience: results from a national survey suggest postoperative pain continues to be undermanaged. Anesth Analg. 2003 Aug;97(2):534-540. doi: 10.1213/01.ANE.0000068822.10113.9E. PMID 12873949
- [Result] Luketich JD, Land SR, Sullivan EA, Alvelo-Rivera M, Ward J, Buenaventura PO, Landreneau RJ, Hart LA, Fernando HC. Thoracic epidural versus intercostal nerve catheter plus patient-controlled analgesia: a randomized study. Ann Thorac Surg. 2005 Jun;79(6):1845-9; discussion 1849-50. doi: 10.1016/j.athoracsur.2004.10.055. PMID 15919269
- [Result] Oderda GM, Said Q, Evans RS, Stoddard GJ, Lloyd J, Jackson K, Rublee D, Samore MH. Opioid-related adverse drug events in surgical hospitalizations: impact on costs and length of stay. Ann Pharmacother. 2007 Mar;41(3):400-6. doi: 10.1345/aph.1H386. Epub 2007 Mar 6. PMID 17341537
- [Result] Richard BM, Rickert DE, Newton PE, Ott LR, Haan D, Brubaker AN, Cole PI, Ross PE, Rebelatto MC, Nelson KG. Safety Evaluation of EXPAREL (DepoFoam Bupivacaine) Administered by Repeated Subcutaneous Injection in Rabbits and Dogs: Species Comparison. J Drug Deliv. 2011;2011:467429. doi: 10.1155/2011/467429. Epub 2011 Oct 5. PMID 22013534
- [Result] American Society of Anesthesiologists Task Force on Acute Pain Management. Practice guidelines for acute pain management in the perioperative setting: an updated report by the American Society of Anesthesiologists Task Force on Acute Pain Management. Anesthesiology. 2012 Feb;116(2):248-73. doi: 10.1097/ALN.0b013e31823c1030. No abstract available. PMID 22227789
- [Result] Chahar P, Cummings KC 3rd. Liposomal bupivacaine: a review of a new bupivacaine formulation. J Pain Res. 2012;5:257-64. doi: 10.2147/JPR.S27894. Epub 2012 Aug 14. PMID 23049275
- [Result] Golembiewski J, Dasta J. Evolving Role of Local Anesthetics in Managing Postsurgical Analgesia. Clin Ther. 2015 Jun 1;37(6):1354-71. doi: 10.1016/j.clinthera.2015.03.017. Epub 2015 Apr 10. PMID 25866297
- [Result] Kelly MA. Current Postoperative Pain Management Protocols Contribute to the Opioid Epidemic in the United States. Am J Orthop (Belle Mead NJ). 2015 Oct;44(10 Suppl):S5-8. PMID 26447431
- [Result] Khalil KG, Boutrous ML, Irani AD, Miller CC 3rd, Pawelek TR, Estrera AL, Safi HJ. Operative Intercostal Nerve Blocks With Long-Acting Bupivacaine Liposome for Pain Control After Thoracotomy. Ann Thorac Surg. 2015 Dec;100(6):2013-8. doi: 10.1016/j.athoracsur.2015.08.017. Epub 2015 Oct 24. PMID 26507422
- [Result] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739
- [Result] Uskova A, O'Connor JE. Liposomal bupivacaine for regional anesthesia. Curr Opin Anaesthesiol. 2015 Oct;28(5):593-7. doi: 10.1097/ACO.0000000000000240. PMID 26308513
- [Result] Biswas S, Verma R, Bhatia VK, Chaudhary AK, Chandra G, Prakash R. Comparison between Thoracic Epidural Block and Thoracic Paravertebral Block for Post Thoracotomy Pain Relief. J Clin Diagn Res. 2016 Sep;10(9):UC08-UC12. doi: 10.7860/JCDR/2016/19159.8489. Epub 2016 Sep 1. PMID 27790554 (Retraction: PMID 32662777 J Clin Diagn Res. 2020 Jul;14(7):ZZ01)
- [Result] Redan JA, Wells T, Reeder S, McCarus SD. Reducing Opioid Adverse Events: A Safe Way to Improve Outcomes. Surg Technol Int. 2016 Apr;28:101-9. PMID 27042786
- [Result] Clinicians' quick reference guide to postoperative pain management in adults. Pain Management Guideline Panel. Agency for Health Care Policy and Research, US Department of Health and Human Services. J Pain Symptom Manage. 1992 May;7(4):214-28. PMID 1517644
- See also: HCAHPS (Hospital Consumer Assessment of Healthcare Providers and Systems) fact sheet — http://www.hcahpsonline.org/Files/HCAHPS_Fact_Sheet_June_2015.pdf